CLINICAL TRIAL: NCT00385320
Title: To Assess the Efficacy, Immuno & Safety of 2 Doses of GSK HRV Vaccine at Different Virus Concentrations in Healthy Infants Aged 2 Months & Previously Uninfected With HRV, Concurrently Given With DTPw-HBV, Hib.
Brief Title: Evaluate Protective Efficacy of Diff Strengths of Human Rotavirus Vaccine After Admn of 2 Doses to Infants Aged 2 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444563/006
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: HRV vaccine

SUMMARY:
The purpose of this study is to test how infants respond to different strengths of the human rotavirus vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infant between, and including, 6 and 12 weeks of age born after a gestation period of 36 to 42 weeks or a birth weight of >2000g.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* Planned administration of oral polio vaccine during the period starting from 2 weeks before each dose of study vaccine(s) and ending 2 weeks after.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* History of diphtheria, tetanus, pertussis, Hib disease and/ or hepatitis B.
* Previous vaccination against diphtheria, tetanus, pertussis, and/or Haemophilus influenzae type b.
* History of allergic disease
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract or other serious medical condition as determined by the investigator.
* Gastroenteritis within 7 days preceding the study vaccine administration (warrants deferral of the vaccination)
* Previous confirmed occurrence of RV GE.
* Household contact with an immunosuppressed individual or pregnant women.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2640 (Actual)
Dates: Start 2001-05-31 (Actual); Primary Completion 2003-04-30 (Actual); Study Completion 2003-04-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of RV GE

SECONDARY OUTCOMES:
Serum RV IgA antibody titre, Viral shedding, Seroprotection/seropositivity status for DTPwHBVHib antigens, Solicited, unsolicited & SAE

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=3349

REFERENCES:
- [Background] Araujo EC, Clemens SA, Oliveira CS, Justino MC, Rubio P, Gabbay YB, da Silva VB, Mascarenhas JD, Noronha VL, Clemens R, Gusmao RH, Sanchez N, Monteiro TA, Linhares AC. Safety, immunogenicity, and protective efficacy of two doses of RIX4414 live attenuated human rotavirus vaccine in healthy infants. J Pediatr (Rio J). 2007 May-Jun;83(3):217-24. doi: 10.2223/JPED.1600. Epub 2007 Mar 20. PMID 17380232
- [Background] Buyse H, Vinals C, Karkada N, Han HH. The human rotavirus vaccine Rotarix in infants: an integrated analysis of safety and reactogenicity. Hum Vaccin Immunother. 2014;10(1):19-24. doi: 10.4161/hv.26476. Epub 2013 Oct 8. PMID 24047799
- [Background] Cheuvart B, Neuzil KM, Steele AD, Cunliffe N, Madhi SA, Karkada N, Han HH, Vinals C. Association of serum anti-rotavirus immunoglobulin A antibody seropositivity and protection against severe rotavirus gastroenteritis: analysis of clinical trials of human rotavirus vaccine. Hum Vaccin Immunother. 2014;10(2):505-11. doi: 10.4161/hv.27097. Epub 2013 Nov 13. PMID 24240068
- [Background] De Vos B, Vesikari T, Linhares AC, Salinas B, Perez-Schael I, Ruiz-Palacios GM, Guerrero Mde L, Phua KB, Delem A, Hardt K. A rotavirus vaccine for prophylaxis of infants against rotavirus gastroenteritis. Pediatr Infect Dis J. 2004 Oct;23(10 Suppl):S179-82. doi: 10.1097/01.inf.0000142370.16514.4a. PMID 15502699
- [Background] De Vos B, Han HH, Bouckenooghe A, Debrus S, Gillard P, Ward R, Cheuvart B. Live attenuated human rotavirus vaccine, RIX4414, provides clinical protection in infants against rotavirus strains with and without shared G and P genotypes: integrated analysis of randomized controlled trials. Pediatr Infect Dis J. 2009 Apr;28(4):261-6. doi: 10.1097/INF.0b013e3181907177. PMID 19289978
- [Background] Linhares AC, Ruiz-Palacios GM, Guerrero ML, Salinas B, Perez-Schael I, Clemens SA, Innis B, Yarzabal JP, Vespa G, Cervantes Y, Hardt K, De Vos B. A short report on highlights of world-wide development of RIX4414: a Latin American experience. Vaccine. 2006 May 1;24(18):3784-5. doi: 10.1016/j.vaccine.2005.07.027. Epub 2005 Jul 26. PMID 16098636
- [Background] Linhares AC, Verstraeten T, Wolleswinkel-van den Bosch J, Clemens R, Breuer T. Rotavirus serotype G9 is associated with more-severe disease in Latin America. Clin Infect Dis. 2006 Aug 1;43(3):312-4. doi: 10.1086/505493. Epub 2006 Jun 23. PMID 16804845
- [Background] Perez-Schael I, Salinas B, Tomat M, Linhares AC, Guerrero ML, Ruiz-Palacios GM, Bouckenooghe A, Yarzabal JP. Efficacy of the human rotavirus vaccine RIX4414 in malnourished children. J Infect Dis. 2007 Aug 15;196(4):537-40. doi: 10.1086/519687. Epub 2007 Jun 29. PMID 17624838
- [Background] Ruiz-Palacios GM, Guerrero ML, Bautista-Marquez A, Ortega-Gallegos H, Tuz-Dzib F, Reyes-Gonzalez L, Rosales-Pedraza G, Martinez-Lopez J, Castanon-Acosta E, Cervantes Y, Costa-Clemens S, DeVos B. Dose response and efficacy of a live, attenuated human rotavirus vaccine in Mexican infants. Pediatrics. 2007 Aug;120(2):e253-61. doi: 10.1542/peds.2006-2630. Epub 2007 Jul 2. PMID 17606534
- [Background] Salinas B, Perez Schael I, Linhares AC, Ruiz Palacios GM, Guerrero ML, Yarzabal JP, Cervantes Y, Costa Clemens S, Damaso S, Hardt K, De Vos B. Evaluation of safety, immunogenicity and efficacy of an attenuated rotavirus vaccine, RIX4414: A randomized, placebo-controlled trial in Latin American infants. Pediatr Infect Dis J. 2005 Sep;24(9):807-16. doi: 10.1097/01.inf.0000178294.13954.a1. PMID 16148848
- [Background] Soriano-Gabarró M et al. (2008) Potential impact of Rotarix according to rotavirus type distribution. Pediatr Infect Dis J. 27(1) Supplement: S28-S32.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 444563/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register